CLINICAL TRIAL: NCT03029091
Title: A Preliminary Open-Label Trial of Losartan Potassium in Participants With Eosinophilic Esophagitis (EoE) With or Without a Connective Tissue Disorder
Brief Title: An Open-Label Trial of Losartan Potassium in Participants With Eosinophilic Esophagitis (EoE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Office of Rare Diseases (ORD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-9021; U54AI117804 (NIH)
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-07

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Losartan

STUDY DESIGN:
Intervention Model Description: This study is an open-label study which means that all participants receive the study medicine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EoE +/- CTD (Experimental): Participants with EoE with and without CTD receive Losartan Potassium, 0.7 - 0.9 mg/kg (titration)/1.0 - 1.4 mg/kg (maintenance) daily for 16 weeks
  Interventions: Drug: Losartan Potassium
- EoE + CTD (Experimental): Participants with EoE with CTD receive Losartan Potassium, 0.7 - 0.9 mg/kg (titration)/1.0 - 1.4 mg/kg (maintenance) daily for 16 weeks
  Interventions: Drug: Losartan Potassium
- EoE - CTD (Experimental): Participants with EoE without CTD receive Losartan Potassium, 0.7 - 0.9 mg/kg (titration)/1.0 - 1.4 mg/kg (maintenance) daily for 16 weeks
  Interventions: Drug: Losartan Potassium

INTERVENTIONS:
Drug: Losartan Potassium — Losartan potassium
  Other Names: Losartan

SUMMARY:
The purpose of this study is to test the safety and effectiveness of Losartan potassium in subjects with eosinophilic esophagitis (EoE) including those with a connective tissue disorder (CTD) and those without a CTD.

DETAILED DESCRIPTION:
The purpose of this research study is to test the safety and effects (good and bad) of Losartan potassium on participants with eosinophilic esophagitis (EoE). If a participant has a connective tissue disorder (CTD) the researchers want to see what effects (good or bad) Losartan has on EoE.

EoE is an inflammatory disease of the esophagus that is typically triggered by exposure to food. Connective tissue disorders (CTDs) are disorders that affect the connective tissues in the body such as tendons and ligaments.

A protein called transforming growth factor (TGF)-beta is associated with both EoE and CTD. Losartan may decrease the amount of TGF-beta and therefore help EoE and CTD.

Losartan is a drug that is approved by the United States Food and Drug Administration (FDA) for use in adults and children over 6 years of age who have high blood pressure. This medication has not been studied in people with EoE.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent
* Confirmed, active EoE (at Screening or within 12 weeks prior to enrollment)
* Does or does not have diagnosis of a connective tissue disorder (CTD)
* Has been on a high dose of proton pump inhibitor (PPI) for at least 8 weeks prior to a diagnostic endoscopy of EoE without histologic resolution (i.e., ≥ 15 eosinophils/HPF).
* Maintain the same diet, swallowed steroid and PPI therapies throughout the duration of the study
* Female participants must be either:

  1. Of non-childbearing potential (pre-menarchal or surgically sterile with documentation). OR
  2. Have a negative urine pregnancy test at screening and at each monthly study visit.

Exclusion Criteria:

* Any past or planned cardiac surgery.
* An aortic root Z-score ≥ 3.0 on a previous echocardiogram.
* Intolerance to Losartan
* A mean blood pressure measurement (both systolic and diastolic) at screening that is below the 2nd percentile for his/her age
* Renal dysfunction
* Another disorder that causes esophageal eosinophilia (e.g., hypereosinophilic syndrome, Churg Strauss vasculitis, eosinophilic granuloma, or a parasitic infection).
* A diagnosis of hepatic insufficiency (e.g., liver failure, history of liver transplantation or persistent liver transaminase elevation).
* A history of abnormal gastric or duodenal biopsy or documented gastrointestinal disorders (e.g., Celiac Disease, Crohn's disease or Helicobacter pylori infection), not including chronic gastritis, chronic duodenitis, mucosal eosinophilia or other eosinophilic gastrointestinal disorders (EGIDs).
* Use of anti-immunoglobulin (Ig)E monoclonal antibody (mAb), anti-tumor necrosis factor (TNF) mAb, anti-IL-5 agents, or anti-IL-13 within 6 months prior to study entry
* Use of methotrexate, cyclosporine, interferon α, or other systemic immunosuppressive or immunomodulating agents within 3 months prior to the screening visit.
* A stricture during endoscopy procedure that prevents passage of the endoscope
* Taking or is planning to take an angiotensin receptor blocker (ARB), angiotensin-converting enzyme inhibitor (ACEI), beta blocker (BB), or calcium-channel blocker therapy at the screening visit or at any time during the study or has been taking any of these medications for 3 months prior to the screening visit.
* Taking or planning to take hydrochlorothiazide, digoxin, warfarin, cimetidine, phenobarbital, rifampin, or fluconazole.
* Taking or planning to take potassium supplements or salt substitutes containing potassium.
* A female participant who is pregnant or nursing or, if of childbearing potential, is not using a medically accepted, effective method of birth control (e.g., condom, oral/injectable/subcutaneous contraceptive, intrauterine device, or sexual abstinence).
* Participated/participating in any investigative drug or device study within 30 days prior to study entry.
* Participated/participating in any investigative biologics study within 3 months prior to study entry.
* Unable to be confirmed, active EoE (at Screening or within 12 weeks prior to enrollment)

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc E Rothenberg, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - University of California, San Diego, La Jolla, California
  - Northwestern University, Chicago, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study information on the Consortium for Eosinophilic Gastrointestinal Disorders (CEGIR) website — https://www.rarediseasesnetwork.org/cms/CEGIR

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from eosinophilic esophagitis specialty clinics (3 sites) in the USA between May 2017 and April 2019.
Pre-assignment Details: 17 participants screened, 2 excluded (2 met exclusion criteria), and 15 initiated the intervention
Groups:
- EoE + CTD: Participants with eosinophilic esophagitis (EoE) with connective tissue disorder (CTD) receive Losartan
- EoE - CTD: Participants with eosinophilic esophagitis (EoE) without connective tissue disorder (CTD) receive Losartan
Period: Overall Study
Arm/Group | EoE + CTD | EoE - CTD
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EoE + CTD | EoE - CTD | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (3.7) | 13.8 (5.0) | 12.0 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 6 | 13
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peak Eosinophil Count
Description: Peak esophageal eosinophil counts were obtained at baseline and 16 weeks. Change in peak eosinophil count is defined as peak count at 16 weeks minus peak count at baseline. A reduction (negative change) in peak count indicates improvement. Peak count is defined as the highest count between the distal and proximal esophageal eosinophil counts.
Time Frame: Baseline, 16 weeks
Population: Per protocol population (protocol violation excluded from data analysis)
Measure: Mean (95% Confidence Interval); unit: eosinophils per high power field
Groups:
- EoE +/- CTD: Participants with eosinophilic esophagitis (EoE) with and without connective tissue disorder (CTD) receive Losartan
Arm/Group | EoE +/- CTD | EoE + CTD | EoE - CTD
Number analyzed (Participants) | 14 | 7 | 7
eosinophils per high power field
  Baseline | 63.3 [41.4 to 85.2] | 67.7 [21.0 to 114.4] | 58.9 [37.5 to 80.2]
  Change | -11.2 [-36.9 to 14.5] | -1.9 [-40.6 to 36.9] | -20.6 [-65.2 to 24.0]

2. Primary Outcome: Number of Serious and Grade 3 or Higher Adverse Events
Description: The occurrence of serious adverse events and Grade 3 and higher adverse events from Week 0 to Week 20
Time Frame: 20 weeks after the start of treatment (16 weeks treatment and 4 weeks follow-up)
Population: Intent to treat analysis including participants enrolled in the study
Measure: Number; unit: events
Arm/Group | EoE +/- CTD | EoE + CTD | EoE - CTD
Number analyzed (Participants) | 15 | 8 | 7
events
  Serious Adverse Events | 0 | 0 | 0
  Grade 3 or higher adverse events | 1 | 0 | 1

3. Secondary Outcome: Percent of Participants in Complete and Partial Histologic Remission at 16 Weeks
Description: Percent of participants in complete and partial histologic remission. Complete remission is defined as esophageal peak eosinophil count ≤ 1 eosinophils per high powered field (eos/hpf). Partial remission is defined as esophageal peak eosinophil count of 2 - 14 eos/hpf.
Time Frame: 16 weeks
Population: Per protocol population (protocol violation excluded from data analysis)
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | EoE +/- CTD | EoE + CTD | EoE - CTD
Number analyzed (Participants) | 14 | 7 | 7
percentage of subjects
  Complete remission (≤ 1 eos/hpf) | 7 [0 to 34] | 14 [0 to 58] | 0 [0 to 41]
  Partial remission (2 - 14 eos/hpf) | 21 [5 to 51] | 14 [0 to 58] | 29 [4 to 71]

4. Secondary Outcome: Change From Baseline in Total Histology Scoring System
Description: The histology scoring system (HSS) measures the severity (grade) and extent (stage) of eight histologic abnormalities in the esophagus including eosinophilic inflammation, eosinophilic abscess, eosinophilic surface layering, surface epithelial alteration, dilated intercellular spaces, basal zone hyperplasia, dyskeratotic epithelial cells, and lamina propria fibrosis. Total score is the sum of grade and stage scores from the esophageal biopsy (distal, mid, or proximal) with the highest score (worst abnormalities) divided by the maximum possible score for the biopsy. Total scores range from 0 - 2 with higher scores indicating worse abnormalities. Histology scores were obtained at baseline and 16 weeks. Change in total histology scoring system (HSS) is defined as total HSS score at 16 weeks minus total HSS score at baseline. A reduction (negative change) in score indicates improvement.
Time Frame: Baseline, 16 weeks
Population: Per protocol population (protocol violation excluded from data analysis).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | EoE +/- CTD | EoE + CTD | EoE - CTD
Number analyzed (Participants) | 14 | 7 | 7
score on a scale
  Baseline - Total HSS | 0.79 [0.65 to 0.93] | 0.89 [0.69 to 1.09] | 0.70 [0.48 to 0.92]
  Change - Total HSS | -0.09 [-0.28 to 0.10] | -0.15 [-0.47 to 0.17] | -0.03 [-0.33 to 0.28]

5. Secondary Outcome: Change From Baseline in Total Endoscopic Reference Score
Description: The endoscopic reference score (EREFS) utilizes standardized criteria for the presence and degree of 5 major endoscopic features (edema, fixed rings, exudates, furrows, strictures). Total score is the sum of the five feature scores from the distal and proximal esophagus. Total scores range from 0 - 18 with higher scores indicating worse features. Endoscopic features were assessed at baseline and 16 weeks. Change in total endoscopic reference score is defined as total score at 16 weeks minus total score at baseline. A reduction (negative change) in score indicates improvement.
Time Frame: Baseline, 16 weeks
Population: Per protocol population (protocol violation excluded from data analysis).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | EoE +/- CTD | EoE + CTD | EoE - CTD
Number analyzed (Participants) | 14 | 7 | 7
score on a scale
  Baseline - EREFS Total Score | 5.1 [3.6 to 6.7] | 5.4 [3.4 to 7.5] | 4.9 [1.9 to 7.9]
  Change - EREFS Total Score | -1.3 [-2.6 to 0.0] | -1.7 [-3.2 to -0.2] | -0.9 [-3.6 to 1.8]

6. Secondary Outcome: Change From Baseline in PEESS V2.0
Description: The Pediatric Eosinophilic Esophagitis Symptom Score (PEESS) V2.0 questionnaire captures EoE-specific symptoms (dysphagia, gastroesophageal reflux, nausea/vomiting, and pain) as reported by their parents (for children 2-18 years of age). The range for PEESS v2.0 scores is 0 to 100, with a higher score being indicative of more frequent and/or severe symptoms. Scores were obtained at baseline and 16 weeks. Change in score is defined as total score at 16 weeks minus total score at baseline as completed by parent proxy.
Time Frame: Baseline,16 weeks
Population: Per protocol population (protocol violation excluded from data analysis)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | EoE +/- CTD | EoE + CTD | EoE - CTD
Number analyzed (Participants) | 13 | 7 | 6
score on a scale
  Baseline - PEESS Total Score | 29.9 [15.5 to 44.4] | 32.7 [6.36 to 59.0] | 26.7 [6.3 to 47.1]
  Change - PEESS Total Score: number analyzed (Participants) | 12 | 6 | 6
  Change - PEESS Total Score | -9.7 [-18.3 to -1.1] | -12.5 [-31.2 to 6.2] | -6.89 [-15.3 to 1.6]

7. Secondary Outcome: Change From Baseline in PedsQL EoE
Description: The Pediatric Eosinophilic Esophagitis Quality of Life Inventory (PedsQL EoE) measures symptoms and problems related to treatment, worry, communication, food/eating, and feelings. The range for PedsQL 3.0 EoE scores is 0 to 100, with a higher score indicating better quality of life. Scores were obtained at baseline and 16 weeks. Change in score is defined as the PedsQL EoE total score at 16 weeks minus total score at baseline as reported by parent proxy.
Time Frame: Baseline, 16 weeks
Population: Per protocol population (protocol violation excluded from data analysis)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | EoE +/- CTD | EoE + CTD | EoE - CTD
Number analyzed (Participants) | 13 | 7 | 6
score on a scale
  Baseline - PedsQL Total Score | 74.4 [64.2 to 84.5] | 73.3 [58.7 to 87.8] | 75.6 [55.3 to 96.0]
  Change - PedsQL Total Score | 6.7 [-0.1 to 13.5] | 4.8 [-7.5 to 17.1] | 9.0 [-0.4 to 18.3]

ADVERSE EVENTS:
Time Frame: From informed consent to 30 days after the cessation of treatment, an average of about 24 weeks
Arm/Group | EoE +/- CTD | EoE + CTD | EoE - CTD
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 12/15 | 7/8 | 5/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EoE +/- CTD (N=15) | EoE + CTD (N=8) | EoE - CTD (N=7)
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0
Upper Respiratory Infection (Infections and infestations) | 2 | 1 | 1
Fever (Infections and infestations) | 1 | 0 | 1
Rhinitis Infective (Infections and infestations) | 1 | 1 | 0
Common Cold (General disorders) | 1 | 0 | 1
Creatinine increased (Investigations) | 2 | 1 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Vasovagal reaction (Nervous system disorders) | 1 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 1
Lightheaded (Social circumstances) | 1 | 0 | 1
Transient Dizziness (General disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT03029091/SAP_000.pdf
  • Study Protocol (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT03029091/Prot_001.pdf